CLINICAL TRIAL: NCT01135966
Title: Resistance Training in Patients With Chronic Obstructive Lung Disease (COPD): Whole Body Vibration Versus Conventional Resistance Training
Acronym: REWORK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/157
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: COPD
Keywords: COPD; Whole Body Vibration training; Conventional resistance training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional training (Active Comparator)
  Interventions: Behavioral: Conventional resistance training program
- Whole body vibration training (Experimental)
  Interventions: Behavioral: Whole body vibration resistance training program

INTERVENTIONS:
Behavioral: Conventional resistance training program — Conventional resistance training program is followed.
  Arms: Conventional training
Behavioral: Whole body vibration resistance training program — WBV training on FITVIBE
  Arms: Whole body vibration training

SUMMARY:
Pulmonary rehabilitation has been emerged as a recommended standard of care for patients with chronic lung disease based on a growing body of scientific evidence. A set of evidence-based guidelines were published in American College of Chest Physicians (ACCP) and the American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR). Since then, the published literature in pulmonary rehabilitation has increased substantially, and other societies have published important statements about pulmonary rehabilitation (eg, the American Thoracic Society and the European Respiratory Society).

In patients with COPD, there is a strong scientific basis for implementing conventional resistance training (CRT) in addition to endurance training. Endurance training, such as walking, is a key component of pulmonary rehabilitation and improves in exercise tolerance and muscular endurance. However, this type of training may not reverse muscle weakness or atrophy. For that reason, strength training seems to be the optimum training modality to increase muscle mass and strength.

Recently, Whole-Body-Vibration (WBV) training has been promoted as an alternative for resistance training on multigym equipment. In WBV training, the subject stands on a platform that generates vertical sinusoidal vibration, during which static and dynamic exercises can be performed.

The present study is conducted to provide an answer on the following question: will a resistance training program, such as the whole body vibration, be even effective than a conventional resistance training program in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD candidate for pulmonary rehabilitation
* Men and female between 40 and 80 years of age
* Written informed consent to participate

Exclusion Criteria:

* Severe cardiac, neurological and orthopedic co-morbidity interfering with exercise training.
* Pacemaker
* Hip, knee of shoulder prosthesis or recently introduced spirals, metal pens, bolts or plates
* Uncontrolled diabetes, epilepsy or migraine
* Osteoporotic or metastatic fractures, acute hernia, discopathy, spondylitis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
estimation of the change of 6 MWD before and after 12 weeks resistance training program (CRT versus WBV training) | before and after 12 weeks
  estimation of the change of 6 MWD (submaximal walking test)after a 12 week conventional resistance training program or after a 12 week whole body vibration training program

SECONDARY OUTCOMES:
changes in muscle strength (quadriceps force)after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by modified Microfet before and after 12 weeks of training.
changes in body composition after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by bioelectrical impedance analysis: Fat Free Mass (FFM)before and after 12 weeks of training.
changes in maximal exercise capacity after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by cyclo-ergospirometry before and after 12 weeks of training
changes in muscle force after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by handgrip force, maximal inspiratory pressure (PImax) and maximal expiratory pressure (PEmax)before and after 12 weeks of training
changes in Quality of life after CRT or after WBV training in patients with COPD | beforer and after 12 weeks
  measured by CRDQ (Chronic Respiratory Disease Questionnaire)before and after 12 weeks of training
changes in Dyspnea scores after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by Chronic Respiratory Disease Questionnaire domain dyspnea (CRDQd) and by the BORG scale before and after 12 weeks of training.
changes in 6MWD and the endurance test on the bicycle after CRT or after WBV training in patients with COPD | before and after 12 weeks
  measured by endurance test on the bicycle (75% Max. Workload)before and after 12 weeks of training. This test will also be repeated after 6 weeks of training.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Derom, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Salhi B, Malfait TJ, Van Maele G, Joos G, van Meerbeeck JP, Derom E. Effects of Whole Body Vibration in Patients With COPD. COPD. 2015;12(5):525-32. doi: 10.3109/15412555.2015.1008693. Epub 2015 Aug 4. PMID 26457458
- See also: website of University Hospital Ghent — http://www.uzgent.be